CLINICAL TRIAL: NCT00331825
Title: A Randomized Controlled Trial Study of Risperidone and Olanzapine for the Schizophrenic Patients With Neuroleptic-Induced Acute Dystonia or Parkinsonism
Brief Title: Risperidone and Olanzapine for the Schizophrenic Patients With Neuroleptic-Induced Acute Dystonia or Parkinsonism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan (Other Government)
Collaborators: Department of Health (Ambiguous)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DOH-890010; TMH-91-01
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2006-05-31 (Estimated); Status verified 2000-02

CONDITIONS: Schizophrenia; Extrapyramidal Syndrome
Keywords: Schizophrenia, EPS, risperidone, olanzapine
MeSH Terms: conditions — Schizophrenia; Basal Ganglia Diseases | interventions — Risperidone; Olanzapine

INTERVENTIONS:
Drug: Risperidone and Olanzapine

SUMMARY:
We initiate a study with research grant from department of health and Taoyuan mental hospital and choose risperidone and olanzapine as study medications. We compare the incidence of using anticholinergic drugs in schizophrenic patients of Han ethnics with neuroleptic-induced acute dystonia or parkinsonism to test the hypothesis that these two medications have different EPS incidence in EPS intolerant population.

DETAILED DESCRIPTION:
Objective: First generation antipsychotics frequently induced extrapyramidal side effects (EPS). Second generation antipsychotics were the choices for EPS intolerant schizophrenic patients. But which one of second generation antipsychotic was the better choice did not have definitive results. We compared risperidone and olanzapine in schizophrenic patients with acute dystonia or parkinsonism side effects and observed the incidence of needing concomitant anticholinergic drugs. We also collected the data of average dose of risperidone and olanzapine to help the dosing strategy guidelines for EPS intolerant schizophrenic patients.

Method: This randomized, rater-blind, parallel group, flexible dose study enrolled patients from Taoyuan Mental Hospital from July 2000 to July 2003. Schizophrenia (DSM-IV) patients who met the research criteria of neuroleptic-induced acute dystonia or parkinsonism research criteria of DSM-IV and greater than moderate severity (>4) of global impression of extrapyramidal syndrome rating scale (ESRS). 70 patients were random assignment to risperidone or olanzapine for 8 weeks. The primary outcome was to compare the incidence of concomitant anticholinergic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-65 y/o;
* Female patients did not have pregnancy plans and must agree to use reliable pregnancy prevention methods if during childbearing age;
* Meet schizophrenia criteria of DSM-IV;
* Fulfill DSM-IV neuroleptic-induced acute dystonia or parkinsonism research criteria, the severity of acute dystonia or parkinsonism was greater than moderate degree (>4) assessed by global impression of Extrapyramidal System Rating Scale (item 43 and 44 of ESRS);
* Patients or legal responsible people agree to join study and sign informed consent

Exclusion Criteria:

* Had other axis I diagnosis of DSM-IV;
* Unstable major systemic diseases;
* Had neurological disorder influenced to EPS assessment;
* Substance abuse or dependence other then coffee or tobacco within 6 months before study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2000-07; Study Completion 2003-07

PRIMARY OUTCOMES:
Percentage of using concomitant anticholinergic drugs

SECONDARY OUTCOMES:
Scores of Rating Scale (Extrapyramidal System Rating Scale, Brief Psychiatric Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yu Chan, M.D., Study Chair — Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan
Locations (1):
- Taoyuan Mental Hospital, Taoyuan District, Taiwan